CLINICAL TRIAL: NCT06694415
Title: Determining Paediatric Usual Values for Hormones Dosages by Mass Spectrometry
Brief Title: Determining Paediatric Usual Values for Hormones Dosages by LC-MS/MS
Acronym: DOSHOMASS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240887; IDRCB-2024-A01634-43 (Other: ANSM)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Control Condition
Keywords: LC-MS/MS; Hormones; Children; Usual values

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum frozen storage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Control individuals below 20 years of age: blood sample with hormone dosages

SUMMARY:
Liquid chromatography coupled with mass spectrometry (LC-MS/MS) is now the method of choice for steroid hormone analysis, as it enables analyses to be carried out on small-volume samples on a wider range of hormones, with improved specificity compared with immunoassays. Hormone assays currently face a twofold problem: on the one hand, immunoassays are highly dependent on the synthesis of antibody kits manufactured by companies with immunotechnology expertise; on the other hand, these immunoassays may require the use of radioactive products for quantification, generating considerable risks for both staff and environment. There are international recommendations from expert societies (World Anti-Doping Agency, Endocrine society) to develop new, more reliable assay methods, such as LC-MS/MS, and to phase out immuno- and radioassay techniques.

However, changing measurement methods requires the development of reference values to maintain and optimize the management of patients.

The aim of this project is therefore to establish usual values in a paediatric population, through collaboration between the clinical departments of the APHP and the METOMICS laboratory, which has mastered the technology.

DETAILED DESCRIPTION:
This is a prospective, multicentric, non-randomized. The study will be uncontrolled, as it will use subjects considered "healthy" to establish reference values.

Recruitment is planned to take place in hospital consultations at recruiting centers belonging to the AP-HP.

During the blood sample prescribed as part of the follow-up consultation, an additional blood tube will be collected after information, consent and inclusion.

The following acts and procedures will be added as part of the research:

* additional tube, respecting the total volume taken according to weight (maximum volume of 2.7mL);
* Routine circuit for sending and receiving the tube to ensure the relevance of standards established in real life.
* A biological collection will be set up. Pseudonymized data will be collected on a secure REDCap database. The source data will be: Recruiting center; Age; Gender; Pubertal stage if available; Results of blood tests carried out by mass spectrometry as part of this research.

The clinical database will be completed by investigators from the Endocrine Functional Explorations Department at Trousseau Hospital and biologists from the METOMICS Department at Saint-Antoine Hospital. Data will not be processed outside the AP-HP. Data will be kept in an active secured database for the duration of the study and up to 2 years after the last publication, and archived for 15 years.

Mass spectrometry analyses will be carried out under the supervision of Pr Antonin Lamazière, Head of the Clinical Metabolomics Department at Hôpital Saint Antoine. Data from these analyses will be stored in the same clinical laboratory and shared only with/between the principal investigator and the study methodologist.

During the research phase, the collection will be stored at the Clinical Metabolomics Department (METOMICS) laboratory, under the responsibility of Prof. Antonin Lamazière, for 2 years. At the end of the research, the samples will be stored for a maximum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≤ 20 years old
* undergoing a blood sample as part of their pathology routine follow-up

Exclusion Criteria:

* Any identified or suspected endocrine pathology
* Any acute infectious or inflammatory disorder

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients followed in paediatrics from birth to 20 years undergoing a blood sample as part of their pathology routine follow-up in one of the identified recruiting centers (see below).
  Patients with no identified or suspected endocrine pathology or no infectious or inflammatory disorder.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
to determine paediatric usual values for hormones dosages by mass spectrometry | 1 week
  internal quality control (IQC) suitability/match between the one provided by the manufacturer or developed in-house, and inter-laboratory comparisons (EQA/EIL)

CONTACTS AND LOCATIONS:
Overall Officials: Eloïse Giabicani, MD, PhD, Principal Investigator — Organizational Affiliation: Assistance Publique - Hôpitaux de Paris (AP-HP en général)
Locations (1):
- Service d'Endocrinologie Pédiatrique-Explorations Fonctionnelles Hôpital Trousseau, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided